CLINICAL TRIAL: NCT00356590
Title: Open-Label Extension Treatment With Etanercept (TNFR:Fc) for Participating Patients in Etanercept (TNFR:Fc) Clinical Trial 016.0012
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20021623; 16.0023
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Etanercept; Long-term Safety; Enbrel
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- 1 (Other)
  Interventions: Biological: Etanercept

INTERVENTIONS:
Biological: Etanercept — Etanercept (TNFR:Fc) will be administered 50 mg per week as two 25 mg subcutaneous injections at separate sites, given either on the same day or 3 or 4 days apart.

SUMMARY:
This is an open label, multicenter study for extended treatment of patients who have participated in the Immunex clinical study 016.0012. The primary objective of this study is to evaluate the long term safety of etanercept (TNFR:Fc) in patients with early stage rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria: - Previous enrollment in Immunex protocol 016.0012.

* No clinically significant adverse events thought to be due to etanercept (TNFR:Fc) during previous treatment.
* Negative serum pregnancy test not more than 14 days before the first dose of study drug in females of childbearing potential.
* No more than one NSAID at a dose not greater than the maximum recommended dose and stable for at least two weeks prior to administration of etanercept (TNFR:Fc). Exclusion Criteria:
* Previous receipt of etanercept (TNFR:Fc) (p55), antibody to TNF, anti-CD4 antibody, or diphtheria IL-2 fusion protein.
* Receipt of investigational drugs or biologics (other than etanercept (TNFR:Fc)) within interval between study drug in 016.0012 and this study.
* Receipt of DMARDs (e.g., hydroxychloroquine, oral or injectable gold, azathioprine, cyclosporin, D-penicillamine, sulfasalazine, minocycline, or leflunomide) other than MTX within two weeks prior to the first dose of etanercept (TNFR:Fc) in this study.
* Receipt of cyclophosphamide within 1 month prior to the first dose of etanercept (TNFR:Fc) in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 1998-12; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Genovese MC, Bathon JM, Fleischmann RM, Moreland LW, Martin RW, Whitmore JB, Tsuji WH, Leff JA. Longterm safety, efficacy, and radiographic outcome with etanercept treatment in patients with early rheumatoid arthritis. J Rheumatol. 2005 Jul;32(7):1232-42. PMID 15996057
- [Result] Genovese MC, Bathon JM, Martin RW, Fleischmann RM, Tesser JR, Schiff MH, Keystone EC, Wasko MC, Moreland LW, Weaver AL, Markenson J, Cannon GW, Spencer-Green G, Finck BK. Etanercept versus methotrexate in patients with early rheumatoid arthritis: two-year radiographic and clinical outcomes. Arthritis Rheum. 2002 Jun;46(6):1443-50. doi: 10.1002/art.10308. PMID 12115173
- [Derived] Weinblatt ME, Bathon JM, Kremer JM, Fleischmann RM, Schiff MH, Martin RW, Baumgartner SW, Park GS, Mancini EL, Genovese MC. Safety and efficacy of etanercept beyond 10 years of therapy in North American patients with early and longstanding rheumatoid arthritis. Arthritis Care Res (Hoboken). 2011 Mar;63(3):373-82. doi: 10.1002/acr.20372. Epub 2010 Oct 18. PMID 20957659
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 3 March 1999 through 17 Mar 2000
Groups:
- Etanercept (Enbrel): Etanercept 50 mg subcutaneous dose weekly
Period: Overall Study
Arm/Group | Etanercept (Enbrel)
Started | 468
Completed | 194
Not Completed | 274
Not completed — Adverse Event | 54
Not completed — Death | 10
Not completed — Lost to Follow-up | 35
Not completed — Physician Decision | 46
Not completed — Withdrawal by Subject | 41
Not completed — Completed month 12 only | 2
Not completed — Protocol issues | 6
Not completed — Response status | 28
Not completed — Other | 52

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Age Continuous [Mean (Standard Deviation); unit: Year] | 51.38 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351
  Male | 117
Race/Ethnicity, Customized [Number; unit: Participant]
  Hispanic or Latino | 25
  White or Caucasian | 407
  Other | 4
  American Indian or Alaska Native | 4
  Asian | 5
  Black or African American | 23
Physician Global Assessment of Disease Status [Mean (Standard Deviation); unit: Units on a scale] — Assessed using a 0 - 10 Likert scale, where 0 = asymptomatic and 10 = severe symptoms
  Units on a scale | 5.32 (2.30)
Participant Global Assessment of Disease Status [Mean (Standard Deviation); unit: Units on a scale] — Assessed using a 0 - 10 Likert scale, where 0 = asymptomatic and 10 = severe symptoms
  Units on a scale | 5.51 (2.27)
Participant Pain Visual Analog Scale [Mean (Standard Deviation); unit: Units on a scale] — Assessed using a 10 cm scale ranging from "no pain" (0 cm) to "severe pain" (10 cm).
  Units on a scale | 5.01 (2.62)
Tender Joint Count [Mean (Standard Deviation); unit: Joints] — Based on up to 71 joints
  Joints | 25.81 (16.71)
Swollen Joint Count [Mean (Standard Deviation); unit: Joints] — Based on up to 68 joints
  Joints | 20.30 (12.60)
Health Assessment Questionnaire Disability Index [Mean (Standard Deviation); unit: Units on a scale] — This index is a weighted average of 24 items, each scored 0 (no difficulty) to 3 (unable to function).
  Units on a scale | 1.30 (0.67)
Physical Component Summary Score from SF-36 [Mean (Standard Deviation); unit: Units on a scale] — Physical Component Summary Score from the Short Form-36 Health Survey. This score has a range of 0 to 100, with higher scores indicating better health.
  Units on a scale | 30.42 (9.69)
Mental Component Summary Score from SF-36 [Mean (Standard Deviation); unit: Units on a scale] — Mental Component Summary Score from the Short Form-36 Health Survey. This score has a range of 0 to 100, with higher scores indicating better health.
  Units on a scale | 48.28 (11.52)
C-Reactive Protein [Mean (Standard Deviation); unit: mg/dL] | 3.28 (4.90)
Duration of Morning Stiffness [Mean (Standard Deviation); unit: Minutes] | 182.24 (286.63)

OUTCOME MEASURES:

1. Primary Outcome: Total Exposure to Etanercept With Gaps
Description: Total participant exposure to etanercept (Enbrel) with gaps, calculated as the sum of the times on treatment for all participants. Gaps of up to 14 days from the last treatment in a previous Etanercept study were ignored in calculating time on treatment.
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Participant-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Participant-years | 2882.50

2. Secondary Outcome: ACR20 Response at Month 3
Description: American College of Rheumatology (ACR) 20, defined as a 20% improvement in both tender and swollen joints (78 joints) and a 20% improvement in 3 of 5 items (physician and patient global assessments, patient pain assessment, patient self-assessed disability, and acute-phase C-reactive protein or erythrocyte sedimentation rate)
Time Frame: Baseline and month 3
Population: All enrolled participants who received at least one dose of etanercept and had available data at month 3
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 450
Participants | 276

3. Primary Outcome: Total Exposure-Adjusted Rate of Malignancies
Description: Exposure-adjusted rate of malignancies, excluding nonmelanoma skin cancers, occurring on study within 30 days of the last dose of etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Malignancies per 100 participant-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Malignancies per 100 participant-years | 1.32

4. Primary Outcome: Total Exposure-Adjusted Rate of Deaths
Description: Rate of deaths within 30 days of the last dose of etanercept, adjusted for total exposure to etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Deaths per 100 participant-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Deaths per 100 participant-years | 0.35

5. Primary Outcome: Total Exposure Adjusted Rate of Serious Infectious Events
Description: Exposure-adjusted rate of serious infectious events (associated with hospitalization or IV antibiotics) occurring on study within 30 days of the last dose of etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Events per 100 participant-years | 2.88

6. Primary Outcome: Total Exposure Adjusted Rate of Lymphomas
Description: Rate of lymphomas occurring on study within 30 days of the last dose of etanercept, adjusted for total exposure to etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Lymphomas per 100 participant-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Lymphomas per 100 participant-years | 0.24

7. Primary Outcome: Malignancy
Description: Occurrence of one or more malignancies within the participant on study within 30 days of the last dose of etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Participants | 31

8. Primary Outcome: Lymphoma
Description: Occurrence of one or more lymphomas on study within 30 days of the last dose of etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Participants | 6

9. Primary Outcome: Serious Infectious Event
Description: Occurrence of one or more serious infectious events within the participant on study within 30 days of the last dose of study medication
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Participants | 51

10. Primary Outcome: Total Exposure Adjusted Rate of Serious Adverse Events
Description: Rate of serious adverse events adjusted to total exposure to etanercept (events / exposure * 100)
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Events per 100 patient-years
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Events per 100 patient-years | 13.84

11. Secondary Outcome: Dosing Period
Description: Duration of etanercept dosing
Time Frame: Up to 8 years
Population: All participants who received at least one dose of etanercept
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Days | 2249.6 (1180.00)

12. Secondary Outcome: ACR20 Response at Month 12
Description: American College of Rheumatology (ACR) 20, defined as a 20% improvement in both tender and swollen joints (78 joints) and a 20% improvement in 3 of 5 items (including physician and patient global assessments), in adults
Time Frame: Baseline and month 12
Population: All enrolled participants who received at least one dose of etanercept and had available data at month 12
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 424
Participants | 262

13. Secondary Outcome: ACR50 Response at Month 12
Description: American College of Rheumatology (ACR) 50, defined as a 50% improvement in both tender and swollen joints (78 joints) and a 50% improvement in 3 of 5 items (including physician and patient global assessments), in adults
Time Frame: Baseline and month 12
Population: All enrolled participants who received at least one dose of etanercept and had available data at month 12
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 424
Participants | 192

14. Secondary Outcome: ACR70 Response at Month 12
Description: American College of Rheumatology (ACR) 70, defined as a 70% improvement in both tender and swollen joints (78 joints) and a 70% improvement in 3 of 5 items (including physician and patient global assessments), in adults
Time Frame: Baseline and month 12
Population: All enrolled participants who received at least one dose of etanercept and had available data at month 12
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 424
Participants | 110

15. Secondary Outcome: Standardized Incidence Rate for All SEER Cancers
Description: Standardized incidence rate for all cancers tracked by the National Cancer Institute's Surveillance Epidemiology and End Results (SEER) system, calculated as the ratio of the observed to expected age- and sex-adjusted incidence rates (per person-year) of cancer. Expected rates were based on 1998-2002 SEER data.
Time Frame: Up to 8 years
Population: All participants who received at least one dose of etanercept
Measure: Mean (95% Confidence Interval); unit: Standardized incidence rate
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Standardized incidence rate | 0.99 [0.67 to 1.42]

16. Secondary Outcome: Percent Improvement in Physician Global Assessment of Disease Status From Baseline to Month 12
Description: Percent improvement in the Physician Global Assessment of disease status from baseline to month 12, assessed using a 0 - 10 Likert scale, where 0 = asymptomatic and 10 = severe symptoms
Time Frame: Baseline and month 12
Population: All enrolled participants who received at least one dose of etanercept and had available data for this outcome measure at baseline and month 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 417
Percent change | 50.07 (58.07)

17. Secondary Outcome: Percent Improvement in Participant Global Assessment of Disease Status From Baseline to Month 12
Description: Percent improvement in the Participant Global Assessment of disease status from baseline to month 12, assessed using a 0 - 10 Likert scale, where 0 = asymptomatic and 10 = severe symptoms
Time Frame: Baseline and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 419
Percent change | 35.46 (60.62)

18. Secondary Outcome: Percent Improvement in Participant Pain Visual Analog Scale From Baseline to Month 12
Description: Percent improvement in the Participant Pain Visual Analog Scale (VAS) from baseline to month 12, using a 10 cm scale ranging from "no pain" (0 cm) to "severe pain" (10 cm).
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 422
Percent change | 30.64 (103.25)

19. Secondary Outcome: Percent Improvement in Tender Joint Count From Baseline to Month 12
Description: Percent improvement in tender joint count (based on up to 71 joints) from baseline to month 12. Tender joints were assessed clinically, and the number of such joints was counted at each time point.
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 417
Percent change | 49.70 (147.16)

20. Secondary Outcome: Percent Improvement in Swollen Joint Count From Baseline to Month 12
Description: Percent improvement in swollen joint count (based on up to 68 joints) from baseline to month 12.
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 412
Percent change | 52.04 (87.97)

21. Secondary Outcome: Percent Improvement in HAQ DI From Baseline to Month 12
Description: Percent improvement in the Health Assessment Questionnaire Disability Index (HAQ DI) from baseline to month 12.
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 420
Percent change | 40.91 (66.09)

22. Secondary Outcome: Percent Improvement in the Physical Component Summary Score for SF-36 From Baseline to Month 12
Description: Percent improvement in the Physical Component Summary Score for the Short Form 36 Health Survey (SF-36) from baseline to month 12. This score has a range of 0 to 100, with higher scores indicating better health.
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 422
Percent change | -39.65 (55.43)

23. Secondary Outcome: Percent Improvement in Mental Component Summary Score of SF-36 From Baseline to Month 12
Description: Percent improvement in the Mental Component Summary Score of the Short Form 36 Health Survey (SF-36) from baseline to month 12. This score has a range of 0 to 100, with higher scores indicating better health.
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 422
Percent change | -12.31 (31.48)

24. Secondary Outcome: Percent Improvement in C-Reactive Protein From Baseline to Month 12
Description: Percent improvement in C-reactive protein from baseline to month 12
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 423
Percent change | 31.57 (132.83)

25. Secondary Outcome: Percent Improvement in Duration of Morning Stiffness From Baseline to Month 12
Description: Percent improvement in the duration of morning stiffness from baseline to month 12
Time Frame: Baseline and month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 411
Percent change | 44.08 (156.20)

26. Primary Outcome: Death
Description: Death of the participant on study up to 30 days after the last dose of etanercept
Time Frame: Up to 8 years
Population: All enrolled participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 468
Participants | 10

27. Secondary Outcome: Change From Baseline to Year 2 in Total Sharp Score
Description: Change from baseline to year 2 in Total Sharp Score. This score has a range of 0 to 398, where 0 = no change and higher scores represent a worsening of joint erosions and joint space narrowing.
Time Frame: Baseline, Year 2
Population: All enrolled participants who received at least one dose of etanercept and had available data for this outcome measure at baseline and year 2
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 274
Units on a scale | 1.17 [-10.10 to 32.72]

28. Secondary Outcome: Change From Baseline to Year 2 in Sharp Score Erosion Subscale
Description: Change from baseline to year 2 in the joint erosion subscale of the Total Sharp Score. This subscale has a range of 0 to 230, where 0 = no change and higher values represent a worsening in joint erosions.
Time Frame: Baseline, Year 2
Population: as for outcome 27
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 274
Units on a scale | 0.54 [-8.08 to 20.83]

29. Secondary Outcome: Change From Baseline to Year 2 in Sharp Score Joint Space Narrowing Subscale
Description: Change from baseline to year 2 in the joint space narrowing subscale of the Total Sharp Score. This subscale has a range of 0 to 168, where 0 = no change and higher values represent a worsening of joint space narrowing.
Time Frame: Baseline, Year 2
Population: as for outcome 27
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Etanercept (Enbrel)
Number analyzed (Participants) | 274
Units on a scale | 0.64 [-5.04 to 16.31]

ADVERSE EVENTS:
Time Frame: Up to 9.57 years
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Enbrel
Serious Adverse Events (participants affected / at risk) | 169/468
Other Adverse Events (participants affected / at risk) | 320/468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (N=468)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 4
Arrhythmia (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 5
Coronary artery disease (Cardiac disorders) | 6
Coronary artery occlusion (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 8
Palpitations (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Cleft palate (Congenital, familial and genetic disorders) | 1
Myxoedema (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Peptic ulcer (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 9
Condition aggravated (General disorders) | 11
Death (General disorders) | 1
Impaired healing (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 5
Cholelithiasis (Hepatobiliary disorders) | 2
Anaphylactic shock (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Abdominal infection (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 6
Bronchitis bacterial (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Cholecystitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Haemophilus sepsis (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 2
Orchitis (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 15
Pneumonia escherichia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 3
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 3
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2
Ulna fracture (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1
Biopsy prostate (Investigations) | 1
Colonoscopy (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 5
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 2
Multiple sclerosis (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 4
Transient ischaemic attack (Nervous system disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Conversion disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 3
IgA nephropathy (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Prostatic disorder (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Cystopexy (Surgical and medical procedures) | 1
Incisional hernia repair (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 4
Shoulder arthroplasty (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Arterial thrombosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (N=468)
Dyspepsia (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 26
Fatigue (General disorders) | 26
Injection site erythema (General disorders) | 51
Injection site pruritus (General disorders) | 26
Injection site swelling (General disorders) | 25
Bronchitis (Infections and infestations) | 49
Cystitis (Infections and infestations) | 27
Influenza (Infections and infestations) | 42
Sinusitis (Infections and infestations) | 91
Upper respiratory tract infection (Infections and infestations) | 106
Headache (Nervous system disorders) | 46
Depression (Psychiatric disorders) | 27
Rash (Skin and subcutaneous tissue disorders) | 36
Hypertension (Vascular disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.